CLINICAL TRIAL: NCT06758726
Title: Mitoxantrone Hydrochloride Liposome Injection Combined With Bu/Cy Conditioning on Acute Myeloid Leukaemia Patients With Intermediate/Adverse Risk Disease or Persistently Positive MRD Undergoing Allogeneic Haematopoietic Stem-cell Transplantation: a Prospective, Single-center, Exploratory Clinical Study
Brief Title: Mitoxantrone Hydrochloride Liposome Combined With BU/Cy Were Used as a Conditioning Regimen for Patients With Intermediate/Adverse Risk or Persistently Positive MRD AML
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024064
Record Dates: First submitted 2024-10-23; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-09

CONDITIONS: AML
Keywords: allo-HSCT; MRD+

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome combined with BU/Cy (Other): Mitoxantrone Hydrochloride Liposome combined with BU/Cy were used as a conditioning regimen for patients with intermediate/adverse risk or persistently positive MRD AML.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome combined with BU/Cy

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome combined with BU/Cy — Mitoxantrone hydrochloride liposome (30 mg/m^2) on day -9, iv Busulfan (3.2mg/kg/d) on day -7~-5, iv Cyclophosphamide (60 mg/kg/d) on day -3~-2, iv

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of a conditioning regimen of Mitoxantrone Hydrochloride Liposome in combination with Bu/Cy (M+Bu/Cy) on acute myeloid leukaemia (AML) patients with intermediate/adverse risk disease or persistently positive MRD undergoing allogeneic haematopoietic stem-cell transplantation (allo-HSCT)

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy and safety of a conditioning regimen of Mitoxantrone Hydrochloride Liposome in combination with Bu/Cy (M+Bu/Cy) on acute myeloid leukaemia (AML) patients with intermediate/adverse risk disease or persistently positive MRD undergoing allogeneic haematopoietic stem-cell transplantation (allo-HSCT Mitoxantrone Hydrochloride Liposome combined with BU/Cy were used as a conditioning regimen for patients with intermediate/adverse risk or persistently positive MRD AML.

Mitoxantrone hydrochloride liposome (30 mg/m^2) on day -9, iv Busulfan (3.2mg/kg/d) on day -7~-5, iv Cyclophosphamide (60 mg/kg/d) on day -3~-2, iv

ELIGIBILITY:
Inclusion Criteria:

* 1.Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.

  2. Age: 18-60 years (including 18 and 60 years) 3. Clinically diagnosed AML, excluding acute promyelocytic leukemia. Patients with at least one or more characteristics can be enrolled:
  1. AML patients with intermediate/adverse risk disease according to 2022 ELN recommendations.
  2. AML patients with persistently positive MRD before allo-HSCT. 4. Physical status score of Eastern Oncology Collaboration Group (ECOG) : 0-2. 5. Negative HIV, HBV and HCV. 6. Before the research procedure begins, an ICF must be signed by the patient himself or a close relative. Considering the patient's condition, if signing the ICF by himself is not beneficial to the treatment of the disease, then the legal guardian or a close relative of the patient sign it.

     Exclusion Criteria:
* 1. Relapsed/refractory AML. 2. Prior therapy with doxorubicin or other anthracyclines, and the cumulative dose of doxorubicin > 360 mg/m^2 (1 mg doxorubicin was equivalent to 2 mg daunorubicin or 0.5 mg idarubicin).

  3. Cardiovascular diseases, including but not limited to:
  1. QTc interval >480 ms or long QTc syndrome in screening;
  2. Complete left bundle branch block, 2 or 3 grade atrioventricular block;
  3. Requiring treatment of serious and uncontrolled arrhythmia;
  4. New York Heart Association (NYHA≥2);
  5. Cardiac ejection fraction (EF) was less than 50%;
  6. Myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other history of arrhythmia or clinically serious pericardial disease that requires treatment within the first 6 months of enrollment, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.

  4. Previous or current occurrence of other malignancies (in addition to non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years).

  5. Subjects are suffering from any other uncontrollable disease (including but not limited to: uncontrolled diabetes and hypertension, and advanced infection).

  6. HIV infection. 7. HBsAg or HBcAb positive, with HBV-DNA≥1x10^3 copies/mL; or HCV-RNA≥1x10^3 copies/mL; 8. Uncontrollable infection, mechanical assisted ventilation or hemodynamic instability at enrollment.

  9. Clinically significant severe liver insufficiency (defined as grade C by Child-Pugh), AST or ALT was 5 times higher than the upper limit of normal (ULN), or serum total bilirubin was 2 times higher than the ULN within 5 days prior to enrollment.

  10. End-stage renal insufficiency was diagnosed with creatinine clearance of less than 10ML/min within 5 days prior to enrollment.

  11. Moderate hepatic insufficiency and moderate renal insufficiency were simultaneously diagnosed (moderate hepatic insufficiency was defined ash grade B by Child-Pug; Moderate renal insufficiency is defined as creatinine clearance of less than 50ML/min).

  12. A history of immediate or delayed allergy to similar drug and excipients of the investigate drug.

  13. Pregnant, lactating female or subjects who refuse to use effective contraception during the study.

  14. With a history of severe neurological or psychiatric illness. 15. Not suitable for this study as decided by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
1 year-relapsed free survival (1y-RFS) | 1YEAR
  RFS was defined as time from achieving remission until disease relapse or disease progression.

SECONDARY OUTCOMES:
1 year-overall survival (1y-OS) | 1YEAR
  OS was defined as time from conditioning treatment until death from any cause.
1 year-non-relapse mortality (1y-NRM) | 1YEAR
  NRM was defined as death from any cause not subsequent to relapse or disease progression.
1 year-cumulative incidence of relapse (1y-CIR) | 1YEAR
  CIR was defined as time from conditioning treatment until relapse or disease progression.
Time of neutrophil and platelet engraftment | 8 weeks
  Neutrophil engraftment was defined as the first of 3 consecutive days with absolute neutrophil counts exceeding 0.5×109 cells per L, and platelet engraftment as the first of 3 consecutive days with absolute platelet counts exceeding 20×109 platelets per L without a platelet transfusion.
Complete response (CR) rate | 1YEAR
  CR rate was defined as bone marrow blasts less than 5% with normal maturation of all cell lines, absence of circulating blasts and blasts with Auer rods, absence of extramedullary disease, and absolute neutrophil count ≥1×109 cells per L, platelet count ≥100×109 platelets per L.
Incidence of adverse events | 14 weeks
  Adverse events were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0) except for GVHD; aGVHD and cGVHD were graded according to published guidelines.
Regimenrelated toxicity (RRT) | 4 weeks
  RRT was assessed within 28 days after transplantation and graded according to Bearman's criteria.